CLINICAL TRIAL: NCT04178538
Title: The Effect of Bone Marrow Aspirate, Demineralized Bone Matrix, and InternalBrace™ on the Outcomes of Anterior Cruciate Ligament Reconstruction in Young Adults; Failure Rates and Return to Play
Brief Title: The Effect of Fertilized ACL Technique on Outcomes of ACL Reconstruction in Young Adults
Acronym: FACL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Marshall University (Other)
Collaborators: Arthrex, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1455859
Record Dates: First submitted 2019-10-17; First posted 2019-11-26 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-04

CONDITIONS: ACL Tear; ACL Injury; Arthroscopy; Anterior Cruciate Ligament Tear
Keywords: Anterior cruciate ligament tear; ACL
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- 25 years and older- ACL recon with DBM, Internal brace (Experimental): Patients in this arm will be 25 years of age and over and receive ACL reconstruction augmented with demineralized bone matrix, bone marrow, and internal brace
  Interventions: Procedure: ACL reconstruction with bone marrow, demineralized bone marix, and internal brace augmentation
- 25 years and older- Standard ACL reconstruction (Active Comparator): Patients in this arm will be 25 years of age and over will receive an allograft All-Inside ACL reconstruction
  Interventions: Procedure: Standard ACL reconstruction with all inside technique
- 24 years and younger- ACL recon with DBM, Internal brace (Experimental): In this arm patients 24 years and under that are skeletally mature, will receive ACL reconstruction with a quad tendon autograft augmented with demineralized bone matrix, bone marrow, and internal brace
  Interventions: Procedure: ACL reconstruction with bone marrow, demineralized bone marix, and internal brace augmentation
- 24 years and younger- Standard ACL reconstruction (Active Comparator): In this arm patients 24 years and under that are skeletally mature, will receive ACL reconstruction with a quad tendon autograft standard all inside technique
  Interventions: Procedure: Standard ACL reconstruction with all inside technique

INTERVENTIONS:
Procedure: ACL reconstruction with bone marrow, demineralized bone marix, and internal brace augmentation — ACL reconstruction with bone marrow, demineralized bone marix, and internal brace augmentation with all inside technique
  Arms: 24 years and younger- ACL recon with DBM, Internal brace; 25 years and older- ACL recon with DBM, Internal brace
Procedure: Standard ACL reconstruction with all inside technique — Standard ACL reconstruction with all inside technique
  Arms: 24 years and younger- Standard ACL reconstruction; 25 years and older- Standard ACL reconstruction

SUMMARY:
A prospective study, with outcomes including re-rupture rate and return to sport will be collected following ACL reconstruction. In keeping with the surgeon's standard practice, patients 24 years and under that are skeletally mature, will receive a quad tendon autograft; patients 25 years of age and over will receive an allograft All-Inside ACL reconstruction. These two cohorts will then be randomized into two groups, one with bone marrow/DBM and InternalBrace augmentation, and one without. The study procedures will involve use of x-rays, MRI, CT scan, and surveys at varying time points to assess radiographic, imaging and clinical outcomes.

DETAILED DESCRIPTION:
Graft re-rupture is one of the major complications and causes of reoperation after anterior cruciate ligament (ACL) reconstruction. This is more common in younger athletes. Based on the recent literature the rate of graft re-rupture is about 6-11%. Even with newer techniques and different types of grafts the re-rupture rates and return to play have not improved significantly. Athletes younger than 25 years old have been found to have a 23% risk of secondary ACL injury either on the contralateral or ipsilateral side after an ACL reconstruction. Therefore, there is a direct need to improve the outcomes of ACL reconstruction especially in younger athletes. This could be accomplished with earlier biologic incorporation of the graft and further protecting the graft during the early postoperative period. Quad tendon all-inside reconstruction is a reproducible technique for younger athletes receiving surgery. For patients over the age of 22, allograft is commonly used. Recently autogenous bone marrow aspirate has shown superior radiographic incorporation when used for osteochondral allograft transplantation in the knee. The bone marrow aspirate has also shown the presence of similar mesenchymal stem cell concentrations when harvested from the proximal tibia compared to when harvested from the iliac crest; providing a useful and safe alternative during knee surgery. This bone marrow aspirate can be combined with demineralized bone matrix (DBM) as a medium for incorporation into a femoral and tibial tunnel during reconstruction of an ACL. Recently, as an augment to the procedure, an ultrahigh-molecular-weight polyethylene/polyester suture tape was used as an InternalBrace for an ACL allograft reconstruction and found to be safe and effective. The hypothesis of this study is that the combination of the InternalBrace and biologic addition of autogenous bone marrow aspirate may provide improved functional outcomes, and reduced failure rates after ACL reconstruction.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be age 14-60 years old.
* Must be skeletally mature (Tanner 4) patients, with an ACL deficient knee who desire to have ACL reconstructive surgery using autograft or allograft augmentation.
* Patients with associated meniscal and chondral pathology (except patients falling into exclusion criteria below) will be included in the study; such pathology will be treated at the time of ACL reconstruction at the discretion of the surgeon, (and such pathology and treatment will be recorded).
* An understanding of the purpose of the study, and have signed the informed consent.
* Able to return for all subsequent study visits

Exclusion Criteria:

* Patients with multi-ligament surgery (MCL, PCL, LCL, PMC, or PLC repair or reconstruction),
* Patients whom have had previous ACL reconstructive surgery on ipsilateral knee.
* Patients who are currently pregnant or nursing.
* Patients who have a current infection at the operative site.
* Any condition or personal issue that the surgeon deems ineffective to the outcome of the study.
* Workmen's compensation cases

Ages: 14 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2023-11-11 (Estimated); Study Completion 2023-11-11 (Estimated)

PRIMARY OUTCOMES:
Changes in X rays | 6 months, 1 year, and 2 years
  AP and lateral radiographs of all patients included in the study will be obtained and assessed for changes over the study duration at specified time periods
Changes in International Knee Documentation score | Pre-Op, 2 weeks, 6 weeks, 12 weeks, 6 months, 1 and 2 years post-operatively
  Measures 3 categories: symptoms, sports activity, and knee function with a sum total 0-100 with 100 score having highest functional state and 0 low functioning.
Changes in Visual analog pain scale | Pre-Op, 2 weeks, 6 weeks, 12 weeks, 6 months, 1 and 2 years post-operatively
  High score 10 means high pain, low score 1 means low pain
Change in Knee Injury and Osteoarthritis Outcome (KOOS) Scores | 6 months, 1 and 2 years post-operatively
  five patient-relevant dimensions are scored separately: Pain (nine items); Symptoms (seven items); ADL Function (17 items); Sport and Recreation Function (five items); Quality of Life (four items). A Likert scale is used and all items have five possible answer options scored from 0 (No problems) to 4 (Extreme problems) and each of the five scores is calculated as the sum of the items included. Scores are transformed to a 0-100 scale, with zero representing extreme knee problems and 100 representing no knee problems
Change in THE VETERANS RAND 12 ITEM HEALTH SURVEY | 6 months, 1 and 2 years post-operatively
  patient-reported global health measure that is used to assess a patient's overall perspective of their health. seven different health domains: general health perceptions, physical functioning, role limitations due to physical and emotional problems, bodily pain, energy/fatigue levels, social functioning and mental health. Answers are summarized into two scores, a Physical Component Score (PCS) and a Mental Component Score (MCS) which then provides an important contrast between the respondents physical and psychological health status. results of the VR-12 are summarized as two scores - a Mental Component Score (MCS) and a Physical Component Score (PCS). The scores may be reported as Z-scores (difference compared to the population average, measured in standard deviations). The United States population average PCS and MCS are both 50 points.
Change in LYSHOLM KNEE QUESTIONNAIRE | 6 months, 1 and 2 years post-operatively
  patient-reported instrument that consists of subscales for pain, instability, locking, swelling, limp, stair climbing, squatting, and the need for support. Scores range from 0 (worse disability) to 100 (less disability).
Change in MARX ACTIVITY SCALE FORM | 6 months, 1 and 2 years post-operatively
  MARX focuses on four activity points: running, deceleration, cutting (changing directions while running), and pivoting. Patients are asked to indicate approximately how many times in the past 12 months they performed each of these activities while at their healthiest and most active state. The four knee functions are rated on a 5-point scale of frequency and scores are added up to a maximum of 16 points with a higher score indicating more frequent participation.
Return to play | Until study completion, average of 1 year
  We will assess the time it takes from date of ACl reconstruction until the patient returs to sporting activiy
graft re-rupture rate | Until study completion, average of 1 year
  We will assess patients for incidence of graft rerupture rate during rehab or after return to play
MRI | 12 weeks post op
  MIR scans will be performed first 6 patients in each group will receive MRIs of the knee to visualize graft maturation.
CT scan of operative knee | 6 months post op
  At six (6) months, the first 6 patients in each group will receive CT scans of the knee to assess tunnel widening

CONTACTS AND LOCATIONS:
Overall Officials: Chad Lavender, MD, Principal Investigator — Marshall University
Locations (1):
- Marshall University Department of Orthopedics, Huntington, West Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Crawford SN, Waterman BR, Lubowitz JH. Long-term failure of anterior cruciate ligament reconstruction. Arthroscopy. 2013 Sep;29(9):1566-71. doi: 10.1016/j.arthro.2013.04.014. Epub 2013 Jun 29. PMID 23820260
- [Background] Wiggins AJ, Grandhi RK, Schneider DK, Stanfield D, Webster KE, Myer GD. Risk of Secondary Injury in Younger Athletes After Anterior Cruciate Ligament Reconstruction: A Systematic Review and Meta-analysis. Am J Sports Med. 2016 Jul;44(7):1861-76. doi: 10.1177/0363546515621554. Epub 2016 Jan 15. PMID 26772611
- [Background] Smith PA, Bley JA. Allograft Anterior Cruciate Ligament Reconstruction Utilizing Internal Brace Augmentation. Arthrosc Tech. 2016 Oct 10;5(5):e1143-e1147. doi: 10.1016/j.eats.2016.06.007. eCollection 2016 Oct. PMID 28224069
- [Background] Narbona-Carceles J, Vaquero J, Suarez-Sancho S, Forriol F, Fernandez-Santos ME. Bone marrow mesenchymal stem cell aspirates from alternative sources: is the knee as good as the iliac crest? Injury. 2014 Oct;45 Suppl 4:S42-7. doi: 10.1016/S0020-1383(14)70009-9. PMID 25384474
- [Background] Oladeji LO, Stannard JP, Cook CR, Kfuri M, Crist BD, Smith MJ, Cook JL. Effects of Autogenous Bone Marrow Aspirate Concentrate on Radiographic Integration of Femoral Condylar Osteochondral Allografts. Am J Sports Med. 2017 Oct;45(12):2797-2803. doi: 10.1177/0363546517715725. Epub 2017 Jul 24. PMID 28737949